CLINICAL TRIAL: NCT05033977
Title: Investigating of Difference Between Center-based Physical Therapy and Home-based Physical Therapy After Platelet Rich Plasm Injection in Women With Knee Osteoarthritis
Brief Title: Center-based Physical Therapy and Home-based Physical Therapy After Platelet Rich Plasm Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HANDE GUNEY, Assoc, Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 2021/049
Record Dates: First submitted 2021-05-31; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Exercise; Platelet rich plasma; muscle strength
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: supervised exercise group home exercise group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Center-based Exercise (Experimental): patients did exercises with a physical therapist in a clinic 3 days and 45 minute in a week for 6 weeks.
  The exercise programe included strenghtening and streching exercises. Strenghtening exercises for lower extremity and streching exercises for hamstrings.
  Interventions: Other: Exercise (center-based)
- Home-based exercise (Experimental): Patients did exercises at home every day and 3 times per day. The exercise programe included strenghtening and streching exercises. Strenghtening exercises for lower extremity and streching exercises for hamstrings.
  Interventions: Other: Exercise (home-based)

INTERVENTIONS:
Other: Exercise (center-based) — Exercise therapy with a physical therapist in a clinic.
  Arms: Center-based Exercise
Other: Exercise (home-based) — Patients did exercises at home every day and 3 times per day.
  Arms: Home-based exercise

SUMMARY:
Osteoarthritis (OA) of the knee is a chronic disease characterized by pain, reduced range of motion, instability and effusion in the joint. Moreover, no study has investigated the effect of Platelet-rich Plasma (PRP) in comparison with that of a placebo injection in the same patient with bilateral knee OA. The purpose of this study was to compare the effectiveness of supervised physiotherapy and home exercises after PRP injection in patients with knee OA. The investigator hypothesized that the supervised physiotherapy program would be more effective in decreasing pain and improving muscle strength, physical function, and quality of life than home exercises following PRP injection in patients with knee OA. A total of 30 patients with complete follow-up to 6 weeks post-intervention; 17 patients randomized to the supervised exercise group and 13 patients randomized to the home exercise group. Subjects were recruited from who had radiographic evidence (Kellgren-Lawrence Grade II-III) of knee OA and ranged from 45 to 70 years of age. Measurements including pain during rest and activity, muscle strength assessment, self-estimated functions of the affected knee and functional performance tests for lower extremity strength were performed.

DETAILED DESCRIPTION:
A total of 30 patients with complete follow-up to 6 weeks post-intervention; 17 patients randomized to the supervised exercise group and 13 patients randomized to the home exercise group. Subjects were recruited from who had radiographic evidence (Kellgren-Lawrence Grade II-III) of knee OA and ranged from 45 to 70 years of age. Measurements including pain during rest and activity, muscle strength assessment, self-estimated functions of the affected knee and functional performance tests for lower extremity strength were performed.

Pain Measurement Visual Analog Scale was used to assess the subjects' pain during rest and activity. A 10 cm line was driven and subjects was wanted to mark the point (0; no pain, 10; worst imaginable pain) as representing the pain during rest and activity.

Muscle Strength Measurement Quadriceps, hamstring muscles and the hip stability isometric test (HipSIT) strength were measured with a hand-held digital dynamometer. Each subject was verbally informed before the test in order to ensure correct movement and subjects were asked to perform submaximal contraction against the evaluator's hand before testing. ''Break test'' technique was performed for the strength measurement. According to this technique, the evaluator gradually overcomes the muscle strength and stops when the joint gives way. The quadriceps muscle strength was measured in a sitting position (Hip 90° flexion, knee extended) with hands crossed across the chest. The hand-held dynamometer was positioned on the anterior surface of the lower leg proximal to the ankle during test. Hamstring muscle group measurement was carried out on prone position (Hip neutral position, knee flexion 90°). The hand-held dynamometer was positioned on the posterior surface of the lower leg proximal to the ankle during test. The HipSIT evaluates the abductor, external rotator and extensor muscles of the hip together. This test was performed in a side-lying position (Hips 45° flexion, knees 90° flexion, heels in contact with the limb tested superior to opposing limb as 20° abduction). The hand-held dynamometer was placed on laterally positioned 5 cm above the knee joint interline during test. Each measurement for each muscle was performed 3 times at 30 sec intervals and the higher value was recorded. There was also a minute interval between muscle groups measurements.

Functional Status The Western Ontario and McMaster Universities (WOMAC) index is a disease specific self-administered test for OA to assess functions of the affected joints. It consists of 24 questions (three subscale; pain (5 questions), stiffness (2 questions) and daily activities (17 questions).

Interventions Each subject was informed about knee OA and daily activities that negatively affect the knee OA. They were also asked to use cold press 3 times (10-15 min) a day for 6 weeks. Supervised physiotherapy group performed exercises 3 times a week for 6 weeks under supervision of a physiotherapist after the first evaluation. The subjects in home exercise group were taught exercises and they were informed to do exercises 3 times a week for 6 weeks. Home exercise group was telephoned to motivate them to do exercise or to find out if they have any problem about the exercises once a week for 6 weeks. The exercise programs for each group consisted of these parts: warm up, strengthening, balance and cool down period. The standard exercises were performed by all of the subjects in each group in order to standardize the exercise procedure. We used OMNI Resistance Exercise Scale for perceived effort to standardize elastic-band (Thera-Band; The Hygenic Corporation, Akron, OH) resistance among subjects. Subjects were asked to do 3 repetitions for each exercise starting with lowest resistance elastic band, and the resistance of the elastic band was increased until it reached 5 on the 11-point scale to determine the appropriate elastic band. Second measurements were performed at the end of 6 weeks, the day of routine doctor control for PRP injection. All assessments were performed by the same physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis
* Patients with PRP injections

Exclusion Criteria:

* have any neurologic disease
* have any oncologic disease
* have any other intraarticular injection last 6 months

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Visuel analogue scale | 6 weeks
  Visual Analog Scale was used to assess the subjects' pain during rest and activity. A 10 cm line was driven and subjects was wanted to mark the point (0; no pain, 10; worst imaginable pain) as representing the pain during rest and activity
Muscle Strenght | 6 weeks
  Quadriceps, hamstring muscles and the hip stability isometric test (HipSIT) strength were measured with a hand-held digital dynamometer. Each subject was verbally informed before the test in order to ensure correct movement and subjects were asked to perform submaximal contraction against the evaluator's hand before testing. ''Break test'' technique was performed for the strength measurement.

SECONDARY OUTCOMES:
Physical Function | 6 weeks
  A 30-sec chair stand test and stair climb test were used to assess physical performance. The subjects were asked to stand up from a chair (height: 43cm) and sit down in 30 sec with their arms folded across the chest during the 30-sec chair stand test. The number of the repetitions were recorded. The subjects were asked to ascend and descend 10 steps (step height 20 cm) at a safe and comfortable pace during the stair climb test. The time (sec) of stair ascend and descend were recorded separately.
Knee Function | 6 weeks
  The Western Ontario and McMaster Universities (WOMAC) index is a disease specific self-administered test for OA to assess functions of the affected joints. It consists of 24 questions (three subscale; pain (5 questions), stiffness (2 questions) and daily activities (17 questions)
Weight | 6 weeks
  participants' weight was measured with a digital scale
Height | 6 weeks
  participants' height was measured with a tape measure
Body mass index (BMI) | 6 weeks
  Body Mass Index was calculated using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Güney Deniz, Assoc.,Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT05033977/Prot_SAP_000.pdf